CLINICAL TRIAL: NCT04865328
Title: Impact of OAB Symptoms on Work, Quality of Life and Treatment-seeking Behavior in Croatia
Brief Title: Impact of OAB Symptoms on Quality of Life in Croatia
Acronym: OAB-CRO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Zagreb (Other)
Responsible Party: Principal Investigator, Mislav Mikuš, MD., University of Zagreb
Other Study IDs: PetrovaGyn
Record Dates: First submitted 2021-04-25; First posted 2021-04-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- OAB group: Group with diagnosed overactive bladder.
  Interventions: Other: Overactive Bladder-Validated 8-question Screener (OAB-V8)

INTERVENTIONS:
Other: Overactive Bladder-Validated 8-question Screener (OAB-V8) — OAB-V8 is an eight-item, self-reported questionnaire that assesses the burden of OAB and the degree of bother caused by the symptoms. Since its development as a subscale of the overactive bladder questionnaire (OAB-q), the OAB-V8 questionnaire has been used to screen for OAB and to assess OAB symptom burden and severity.

SUMMARY:
Overactive bladder (OAB) has a negative impact on the daily activities of affected individuals. OAB affects an estimated 12-17% of adults and has a similar reported prevalence in men and women. It has the potential to impair multiple domains of quality of life, including restriction of social and work life, while also resulting in higher healthcare resource use and costs.

The primary objective of the present study was to evaluate, in a Croatian population reporting symptoms of OAB, the effect on work productivity and treatment behaviors (treatment seeking, receiving treatment, treatment dissatisfaction and treatment discontinuation).

ELIGIBILITY:
Inclusion Criteria:

* consenting adult patients who had an OAB diagnosis by their healthcare practitioner and were about to start mirabegron treatment as part of routine clinical practice were eligible for enrollment.

Exclusion Criteria:

* mixed incontinence where stress incontinence was the predominant symptom (as determined by the investigator)
* severe uncontrolled hypertension (i.e. systolic blood pressure ≥180 mm Hg and/or diastolic blood pressure ≥110 mm Hg)
* anxiety and/or depression
* pregnancy
* women who reported having either a current or previous (within one month) urinary tract infection

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with diagnosed overactive bladder without treatment.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-05-10 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
OAB-V8 score > 8 | At the point of recruitment
  The primary study objective is to investigate the impact of individual LUTS on specific outcomes in the population reporting OAB symptoms. OAB-V8 score.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Hospital Centre Zagreb, Croatia, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No
We have no intention to share IPD.

REFERENCES:
- [Derived] Mikus M, Ostroski M, Beljan P, Karadza M, Dumancic S, Sprem Goldstajn M, Coric M, Kalafatic D, Oreskovic S. Validation of the Croatian Version of the 8-Item Overactive Bladder Questionnaire (OAB-V8). Female Pelvic Med Reconstr Surg. 2021 Nov 1;27(11):e687-e690. doi: 10.1097/SPV.0000000000001098. PMID 34534199